CLINICAL TRIAL: NCT03588104
Title: Evaluation of the POWER2DM Diabetes Self-Management Support System Compared With Usual Care for Patients With Diabetes
Brief Title: "POWER2DM Evaluation Campaign"
Acronym: POWER2DMEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, JKSont, Principal investigator, associate professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P17.280
Record Dates: First submitted 2018-05-28; First posted 2018-07-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Type1 Diabetes Mellitus; Type2 Diabetes Mellitus; Diabetes Mellitus; Health Behavior; Self Efficacy
Keywords: Electronic Health (eHealth)
MeSH Terms: conditions — Diabetes Mellitus; Health Behavior

STUDY DESIGN:
Intervention Model Description: Pragmatic randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POWER2DM support group (Experimental): Participants in this group will receive access to the POWER2DM system as an adjunct to usual care. The participants have three intervention visits in which they will use the Shared Decision Making Dashboard to set self-management goals and will use the Self-Management Support system for trying to reach those goals in the periods after the intervention visits.
  Interventions: Device: POWER2DM system
- Usual care group (Active Comparator): Participants in this group will follow their usual diabetes care with their own diabetes care team.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: POWER2DM system — This system consists of two components: 1) the web-based Shared Decision Making Dashboard, used to set self-management goals together with a health care professional with the use of both short- and long-term predictive computer simulation models, and 2) the POWER2DM Self-Management Support System as a mobile application and webpage, used to support behavioural change in DM self-management. The system is fed with data from an activity tracker, a glucose monitor and manual data entry. Power2DM support will be provided as an adjunct to usual care
  Arms: POWER2DM support group
Other: Usual care — Usual care as given to diabetes patients by the patient's diabetes care team.
  Arms: Usual care group

SUMMARY:
Rationale: Hyperglycaemia is an important cause of long-term macro-and microvascular complications in all patients with diabetes mellitus. However, only a small fraction of the patients with diabetes reaches the set target of glycemic control. Problems with adequate self-management usually underlie problems to maintain glycaemic control. Thus, patients need more support in order to reduce the burden and increase the effectiveness of their diabetes self-management. One way to do this is by using integrated technologies and personalized plans for diabetes care. For this purpose, the POWER2DM support system was developed to give patients insight into their condition and support diabetes patients and their health care professionals in setting and achieving self-management goals using predictive computer model simulations and behavioural action plans.

Objective: To provide proof of concept that POWER2DM is safe and effective in improving glycaemic control, improving behavioural/psychosocial and lifestyle markers, and to assess the cost-effectiveness of the approach and to highlight any potential issues that may impede implementation.

Study design: This is a pragmatic randomised controlled trial with 9 months follow-up in which patients will be randomised 1:1 to either Power2DM support (Power2DM group) or usual care (usual care group). There will be evaluation moments at baseline, after 11 weeks, 22 weeks and 37 weeks.

Study population: 230 patients with diabetes (N=115 type 1 diabetes (T1D), N=115 type 2 diabetes (T2D)) recruited from out-patient clinics in the Netherlands (Leiden University Medical Centre and affiliating teaching hospitals N=115) and Córdoba, Spain (Reina Sofia University Hospital N=115).

Intervention: The POWER2DM support group will receive access to the prototype 2 of the POWER2DM system. This system consists of two components: 1) the web-based Shared Decision Making Dashboard, used to set self-management goals together with a health care professional with the use of both short- and long-term predictive computer simulation models, and 2) the POWER2DM Self-Management Support System as a mobile application and webpage, used to support behavioural change in DM self-management. The system is fed with data from an activity tracker, a glucose monitor and manual data entry.

Main study parameters/endpoints: Change in glucose regulation as measured by %HbA1c before and after the intervention compared between the intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed T2DM or T1DM
* Able to self-monitor and work with computer and smart phone with internet connections (as assessed by researcher)

Exclusion Criteria:

* Severe renal insufficiency (eGFR<30ml/min)
* Serious/severe comorbidity that interferes with diabetes outcomes or diabetes self-management including but not limited to: psychiatric diseases, chronic hepatopathy, active malignancy, chronic obstructive pulmonary disease (COPD), disease of the digestive tract, endocrine disorders, cerebrovascular disease with disability
* For female participants: pregnancy or wanting to become pregnant in the coming 9 months
* Concurrent participation in other clinical trials
* Any other situation in which the investigator identifies a potential risk of not being able to perform the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in glycemic control | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Change in HbA1c before and after the intervention compared between the intervention and control group

SECONDARY OUTCOMES:
Amount hypoglycemia | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Amount of hypoglycemia measured by time spent in hypoglycaemia before and after treatment in the Power2DM group compared to the usual care control group
Hypo unawareness | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Hypo unawareness as measured by Clarke's hypo unawareness questionnaire, before and after treatment in the Power2DM group compared to the usual care control group
Incidence of adverse events | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Incidence of adverse events occurring during the study period including serious hypoglycemic events
Mean blood glucose (MBG) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  As derived from continuous glucose measurements by a flash glucose monitoring (FGM) device
Standard deviation of MBG (SDBG) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  As derived from continuous glucose measurements by a FGM device
Largest amplitude of glycemic excursions (LAGE) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  As derived from continuous glucose measurements by a FGM device
Mean amplitude of glycemic excursions (MAGE) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  As derived from continuous glucose measurements by a FGM device
Absolute means of daily differences (MODD) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  As derived from continuous glucose measurements by a FGM device
Time spent in range | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  As derived from continuous glucose measurements by a FGM device
ADVANCE Cardiovascular risk | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  The ADVANCE Cardiovascular Risk Engine, calculates the risk of major cardiovascular disease in patients with type 2 diabetes for the next 4 years (range 0-100%). This is defined as fatal or non-fatal myocardial infarction, stroke or cardiovascular death.
ADVANCE Kidney disease Risk | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  The ADVANCE Kidney Risk Engine, calculates the risk of new-onset albuminuria and major kidney-related events in patients with type 2 diabetes for the next 5 years (range 0-100%). Major kidney-related events are defined as doubling of serum creatinin to >2.26mg/dL, renal replacement therapy, or renal death.
Major Outcomes T1D | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  The Major Outcomes T1D risk score assess the 3, 5 and 7 year risk of a patient with type 1 diabetes on major outcomes (range 0-100%). These outcomes included major coronary heart disease, stroke, end-stage renal failure, amputations, blindness and all-cause death.
UKPDS risk score | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  The UKPDS risk score calculated the risk a patient with type 2 diabetes will develop coronary heart disease, fatal coronary hear disease, stroke or fatal stroke (range 0-100%)
Q score | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  The Q score is a single metric for a continuous glucose monitoring (CGM) profile which summarize the glucose profile using five factors: central tendency, hyperglycemia, hypoglycemia, intra- and inter daily variations.
Amount of steps | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Average amount of steps per day over a week measured by a step counter
Self-reported exercise time | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Exercise time per week as reported in the POWER2DM system
Frequency of self-monitoring of blood glucose (SMBG) measurements | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Frequency of SMBG measurements as reported by the glucose measurement device
Self-reported adherence to medication plan | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Self-reported adherence to medication plan as reported in the POWER2DM system
Weight | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Weight in kilograms measured on a scale
Body mass index (BMI) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  BMI in kg/m2, computed from height and weight
Diabetes Self-Management Questionnaire Revised (DSMQ-R) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  Subscales: Glucose Management, Dietary Control, Physical Activity, Health Care Use Transformed scale scores can vary between 0-10, with higher scores indicating more effective self-care
Patient utilities by EQ-5D | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  No subscales: EQ-5D provides a general health index with higher scores indicating better general health. QALYs will be calculated from EQ-5D scores.
Problem Areas in Diabetes (PAID) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  The PAID provides a total diabetes distress score (0-100), with higher scores (> 40) indicating more distress.
Mood/Well-being by WHO-5 and Patient Health Questionnaire (PHQ-9) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  WHO-5 provides a total score (0-100) with higher scores indicating better wellbeing, PHQ-9 provides a total score (1-27) indicating a likelihood of depression, with higher scores indicating more depressive symptoms
Technology Acceptance Questionnaire (TAQ) | 5 weeks and 37 weeks
  The TAQ provides scores (1-7) on the following domains: Performance expectancy, Effort expectancy, Social influence, Facilitating conditions, Affect, Self-efficacy, Trust, Motivation and Behavioural intention. Higher scores indicate better acceptance of the system.
Cost-effectiveness | Over 37 weeks
  Costs/quality adjusted life years (QALYs) Costs assessed via cost questionnaire and medication registry. QALYs based on patient utilities measured via EQ5D.
Stress by perceived Stress Scale (PSS) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  The PSS provides a total perceived stress score (0-40), with higher scores indicating more perceived stress.
Patient Assessment of Chronic Illness Care (PACIC) | 0 weeks, 11 weeks, 22 weeks and 37 weeks
  The PACIC measures the patient's perception of the care that they receive.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sont, Ph.D., Principal Investigator — Leiden University Medical Center; Javier Delgado Lista, MD Ph.D., Principal Investigator — Andaluz Health Service
Locations (2):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands
- Reina Sofia University Hospital, Córdoba, Spain

REFERENCES:
- [Derived] Ruissen MM, Torres-Pena JD, Uitbeijerse BS, Arenas de Larriva AP, Huisman SD, Namli T, Salzsieder E, Vogt L, Ploessnig M, van der Putte B, Merle A, Serra G, Rodriguez G, de Graaf AA, de Koning EJP, Delgado-Lista J, Sont JK; POWER2DM Consortium. Clinical impact of an integrated e-health system for diabetes self-management support and shared decision making (POWER2DM): a randomised controlled trial. Diabetologia. 2023 Dec;66(12):2213-2225. doi: 10.1007/s00125-023-06006-2. Epub 2023 Sep 29. PMID 37775611